CLINICAL TRIAL: NCT05619614
Title: The Influence of Artificial Intelligence (AI) Assisted Polyp Detection (Discovery System) on Visual Gaze Patterns During Real-time Colonoscopy
Brief Title: The Influence of Artificial Intelligence (AI )Assisted Polyp Detection (Discovery System) on Visual Gaze Patterns During Real-time Colonoscopy
Acronym: REVEAL
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Utrecht University (Other); Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13870
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-04

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients: Participating patients who undergo colonoscopy
- Endoscopists CADe: Physicians performing CADe colonoscopy
  Interventions: Device: eye-tracking glasses
- Endoscopists CC: Physicians performing conventional colonoscopy
  Interventions: Device: eye-tracking glasses

INTERVENTIONS:
Device: eye-tracking glasses — endoscopists wear eye-tracking glasses during real-time colonoscopy
  Groups: Endoscopists CADe; Endoscopists CC

SUMMARY:
In this study, the investigators aim to assess the influence of a computer-aided detection (CADe) system on the visual gaze patterns of endoscopists in order to further understand the effect of AI during real-time colonoscopy.

ELIGIBILITY:
Inclusion Criteria of patients:

* Referred for diagnostic, screening or surveillance colonoscopy

Exclusion Criteria of patients:

* Therapeutic procedure
* Boston Bowel Prep Score (BBPS) score of <6

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults who are referred for regular care colonoscopy
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Mean gaze time per area of influence | End of colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center Nijmegen, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No